CLINICAL TRIAL: NCT00812812
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group , Flexible Dose Study to Evaluate the Efficacy and Safety of Paxil® Tablets in Children and Adolescents With Major Depressive Disorder<Post-marketing Clinical Study>
Brief Title: Paxil Japanese Post Marketing Paediatric Study in Depression (Double-blind, Placebo Controlled Study)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 112487
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2011-10-13 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Depressive Disorder
Keywords: paroxetine; selective serotonin reuptake inhibitor; CDRS-R; children and adolescents
MeSH Terms: conditions — Depressive Disorder | interventions — Paroxetine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paroxetine group (Experimental): paroxetine 10-40mg/day
  Interventions: Drug: paroxetine 10mg tablet; Drug: paroxetine 20mg tablet; Drug: matched placebo to paroxetine 10mg; Drug: matched placebo to paroxetine 20mg
- placebo group (Placebo Comparator): matched placebo to paroxetine
  Interventions: Drug: matched placebo to paroxetine 10mg; Drug: matched placebo to paroxetine 20mg

INTERVENTIONS:
Drug: paroxetine 10mg tablet — 1 or 2 tablet(s) once a day
  Other Names: Paxil
  Arms: paroxetine group
Drug: paroxetine 20mg tablet — 1 tablet once a day
  Other Names: Paxil
  Arms: paroxetine group
Drug: matched placebo to paroxetine 10mg — 2 tablets once a day
Drug: matched placebo to paroxetine 20mg — 1 tablet once a day

SUMMARY:
This study is designed to compare the efficacy of oral paroxetine 10 to 40 mg/day (initial dose:10 mg/day) versus placebo administered once daily (after evening meal) for 8 weeks in children and adolescents with major depressive disorder (MDD) based on the change from baseline to Week 8/end-of-study in the CDRS-R total score in a randomized, double-blind, placebo-controlled parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

run-in period: A subject will be considered eligible for the study only if all of the following criteria apply at start of placebo run-in period.

* Patients who are diagnosed with the following depressive disorders according to the DSM-IV-TR criteria, and currently presents with a depressive episodes. Depressive disorders: MDD, single episode (296.2), MDD, recurrent (296.3)
* 7 years and older and under 18 years old (at the time of consent obtained)
* Patients with a total raw summary score on the CDRS-R of 45 or greater at the Week -2 visit.
* Patients whose legally acceptable representative (e.g., caretaker, custodian) is able to give written consent to participation to this study. Patients aged 12 and above at the time of consent obtained should be able to sign the informed consent on one's own. Efforts should be exerted in obtaining the informed assent in writing from patients aged less than 12.
* Patients with ideal body weight +/- 2SD
* Gender: Male or female

treatment period:

Subjects who meet the following criteria at Week 0 (Baseline) may be progressed to the Treatment period:

- Patients with a total raw summary score on the CDRS-R at Week 0 visit of 45 or greater.

Exclusion Criteria

run-in period:

A subject will not be eligible for inclusion to this study if any of the following criteria applies at start of run-in period:

* Patients who in the investigator's judgment presented with a clinically predominant Axis I disorder other than MDD (e.g. dysthymic disorder, eating disorders, Specific phobia, PTSD, OCD, Panic disorder, etc)
* Patients with any history of a psychotic episode or psychotic disorder (including schizophrenia ), or complication of these diseases.
* Patients with a history of a bipolar disorder, or complication of these diseases.
* Patients with Attention-Deficit, or Hyperactivity Disorder
* Patients with Mental Retardation or Pervasive Development Disorder
* Patients diagnosed with Substance Abuse or Dependence within 12 weeks prior to the Screening visit
* Patients with past treatment experience with the investigational drug (i.e. paroxetine)
* Patients treated with electroconvulsive therapy in the immediate 12 weeks prior to the Screening visit
* Patients with past history of serotonin syndrome and neuroleptic malignant syndrome.
* Patients with CDRS-R score of "suicidal ideation" of 3 or greater. Or patients whose C-SSRS assessment suggests that they are or have been at significant risk for harming themselves or have actually harmed themselves, or who, in the opinion of the chief investigator (subinvestigator), are at significant risk for harming self.
* Patients with past history of suicide attempt, self harm(excluding "no suicidal intent " ), or an intentional overdose (excluding obviously unintentional overdose)
* Patients who have been treated with other clinical trial investigational drug (including post-marketing clinical trial) in the immediate past 3 months of the Week -2 visit.
* Patients who have taken antidepressant medication 1 week prior to screening.
* Patients with complicated disease of glaucoma.
* Patients with convulsive disorders such as epilepsy or past history of these diseases.
* Patients regularly using drugs (e.g. NSAIDs) that would increase the risk of haemorrhage, or patients with bleeding tendency or haemorrhagic diathesis.
* Patients with severe renal and hepatic disorder.
* Patients with serious organic disorder in the brain.
* Patients with chronic hepatitis type B and/or C which is positive of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibody.
* Patients with a current history of carcinoma or malignant tumor, or complication of these diseases.
* Female patients who are pregnant, lactating, or who might be pregnant, or who wish to be pregnant during the study period
* Patients in the opinion of the chief investigator (subinvestigator) judged as not eligible for the study.
* Patients with clinical significant comorbid impulsivity symptoms.(e.g. Personality Disorder, Conduct Disorder)

treatment period: Subjects for whom any of the following categories apply at Week 0 (start of the treatment period) will not be progressed to the treatment phase.

* Patients with CDRS-R score of "suicidal ideation" of 3 or greater, or patients who, in the opinion of the chief investigator (sub investigator), are at significant risk for harming self
* Patients with variation of the CDRS-R total raw summary score at Week 0 of +/-25% or greater compared to that of Week -2.
* Patients with drug compliance of Drug 1 (run-in placebo) from Week -2 to Week 0 less than 80%.
* Patients, in the opinion of the chief investigator (sub investigator) judged as not appropriate for the study.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Japan (16):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ishikawa
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokushima
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary with a conclusion.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112487 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 3 phases: a 2-week placebo run-in phase, an 8-week treatment phase, and a 0- to 3-week taper phase. In the run-in phase, placebo was administered once daily for 2 weeks. In the treatment phase, paroxetine or placebo was orally administered once daily for 8 weeks. In the taper phase, the dose was gradually reduced.
Groups:
- Placebo: Participants took placebo once daily in the treatment phase (8 weeks) and the taper phase (0 to 3 weeks).
- Paroxetine: Paroxetine at the initial dose of 10 milligrams (mg) was orally administered once daily for the first 2 weeks of the treatment phase (total of 8 weeks). During the next 6 weeks, paroxetine 10 to 20 mg for participants aged 7 to 11 years or 10 to 40 mg for participants aged 12 to 17 years was orally administered. The dose was up-titrated by one level at a time (an increment of 10 mg/day) at intervals of at least 2 weeks based on clinical judgment. During the taper phase, (0 to 3 weeks), the last dose level in the treatment phase was reduced by 10 mg/day at intervals of 1 week to the final dose level of 10 mg/day.
Period: Overall Study
Arm/Group | Placebo | Paroxetine
Started | 27 | 29
Completed | 24 | 25
Not Completed | 3 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Paroxetine: Paroxetine at the initial dose of 10 milligrams (mg) was orally administered once daily for the first 2 weeks of the treatment phase. In the next 6 weeks, paroxetine 10 to 20 mg for participants aged 7 to 11 years or 10 to 40 mg for participants aged 12 to 17 years was orally administered. The dose was up-titrated by one level at a time (an increment of 10 mg/day) at intervals of at least 2 weeks based on clinical judgment. During the taper phase (0 to 3 weeks), the last dose level in the treatment phase was reduced by 10 mg/day at intervals of 1 week to the final dose level of 10 mg/day.
- Total: Total of all reporting groups
Arm/Group | Placebo | Paroxetine | Total
Number analyzed (Participants) | 27 | 29 | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.8 (2.62) | 14.4 (1.99) | 14.6 (2.30)
Gender [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 9 | 13 | 22
Race/Ethnicity, Customized [Number; unit: participants] | 27 | 29 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Children's Depression Rating Scale -Revised (CDRS-R) Total Score at Week 8
Description: The CDRS-R has been widely used for the evaluation of children and adolescents with major depressive disorder (MDD). The CDRS-R total score is the sum of the responses to 17 questions. Each question is graded on a 5- or 7-point scale. The highest possible score is 113 (the most severe measure of depression), and the lowest is 17 (not suffering from depression). CDRS-R scores were assessed by the investigator. The change from Baseline in the CDRS-R total score was calculated as the total score at Week 8 minus the total score at Baseline. The data were adjusted with the total score at Baseline.
Time Frame: Baseline and Week 8
Population: Full Analysis Set (FAS): all participants who entered the treatment phase, but excluding participants without the target indication, participants who received no tablet of the treatment phase medication, or participants who had no post-baseline CDRS-R data. The analysis was performed on the last observation carried forward (LOCF) dataset.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Paroxetine
Number analyzed (Participants) | 27 | 29
scores on a scale | -11.9 (2.54) | -16.5 (2.45)
Statistical Analysis 1: Comparison: Placebo vs Paroxetine; Test type: Superiority or Other; p = 0.198, ANCOVA; Mean Difference (Net) = -4.6, 95% CI 2-sided [-11.7 to 2.5] — Mean difference was estimated as paroxetine minus placebo

2. Secondary Outcome: Change From Baseline in the CDRS-R Total Score at Weeks 1, 2, 3, 4, and 6
Description: as for outcome 1
Time Frame: Baseline and Weeks 1, 2, 3, 4, and 6
Population: FAS. The analysis was performed on the observed case (OC) dataset. Participants whose observation was missing at a particular visit were not included in the analysis for that week.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Paroxetine: Paroxetine at the initial dose of 10 mg was orally administered once daily for the first 2 weeks of the treatment phase. In the next 6 weeks, paroxetine 10 to 20 mg for participants aged 7 to 11 years or 10 to 40 mg for participants aged 12 to 17 years was orally administered. The dose was up-titrated by one level at a time (an increment of 10 mg/day) at intervals of at least 2 weeks based on clinical judgment. During the taper phase (0 to 3 weeks), the last dose level in the treatment phase was reduced by 10 mg/day at intervals of 1 week to the final dose level of 10 mg/day.
Arm/Group | Placebo | Paroxetine
Number analyzed (Participants) | 27 | 29
scores on a scale
  Week 1, n=27, 29 | -4.6 (1.10) | -5.4 (1.06)
  Week 2, n=26, 29 | -4.9 (1.56) | -8.8 (1.48)
  Week 3, n=24, 28 | -10.6 (1.90) | -12.0 (1.76)
  Week 4, n=25, 27 | -12.5 (2.24) | -14.6 (2.15)
  Week 6, n=24, 26 | -14.2 (2.21) | -15.7 (2.12)

3. Secondary Outcome: Number of Clinical Global Impression - Global Improvement (CGI-GI) Responders at Weeks 1, 2, 3, 4, 6, and 8
Description: CGI-GI is assessed on an 8-grade scale: 0, not assessed; 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; and 7, very much worse. CGI-GI was assessed by the investigator. Participants who were rated as 1 (very much improved) or 2 (much improved) were categorized as CGI-GI responders.
Time Frame: Weeks 1, 2, 3, 4, 6, and 8
Population: FAS. The analysis was performed on the OC dataset. Participants whose observation was missing at a particular visit were not included in the analysis for that week. The analysis of data at Week 8 was also performed on the LOCF dataset.
Measure: Number; unit: participants
Arm/Group | Placebo | Paroxetine
Number analyzed (Participants) | 27 | 29
participants
  Week 1, n=27, 29 | 4 | 4
  Week 2, n=26, 29 | 4 | 7
  Week 3, n=24, 28 | 7 | 9
  Week 4, n=25, 27 | 13 | 12
  Week 6, n=24, 26 | 12 | 13
  Week 8 (OC), n=24, 25 | 11 | 14
  Week 8 (LOCF), n=27, 29 | 11 | 15

4. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity of Illness (CGI-SI) Score at Weeks 1, 2, 3, 4, 6, and 8
Description: CGI-SI is assessed on an 8-grade scale: 0, not assessed; 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; and 7, among the most extremely ill. CGI-SI was assessed by the investigator. The change from Baseline in CGI-SI score was calculated as the score at Weeks 1, 2, 3, 4, 6, and 8 minus the score at Baseline.
Time Frame: Baseline and Weeks 1, 2, 3, 4, 6, and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Paroxetine
Number analyzed (Participants) | 27 | 29
scores on a scale
  Week 1, n=27, 29 | -0.1 (0.32) | -0.2 (0.41)
  Week 2, n=26, 29 | -0.1 (0.48) | -0.5 (0.69)
  Week 3, n=24, 28 | -0.3 (0.62) | -0.6 (0.57)
  Week 4, n=25, 27 | -0.5 (0.82) | -0.7 (0.76)
  Week 6, n=24, 26 | -0.5 (0.66) | -0.8 (0.82)
  Week 8 (OC), n=24, 25 | -0.5 (0.72) | -1.0 (0.89)
  Week 8 (LOCF), n=27, 29 | -0.4 (0.75) | -0.9 (0.88)

5. Secondary Outcome: Plasma Paroxetine Concentrations at 12 Hours and 24 Hours After Administration of Study Drug at Week 8 or Withdrawal
Description: Summary statistics for the plasma paroxetine concentrations at each time point were calculated by the dosage just before blood sampling using data from participants in whom plasma samples were collected at either 12 hours (plus or minus 2 hours) or 24 hours (plus or minus 2 hours) after the last administration of the study drug at Week 8 or Withdrawal (up to Week 8).
Time Frame: Week 8 or Withdrawal (up to Week 8)
Population: All participants who received paroxetine and in whom plasma samples were collected at either 12 hours (plus or minus 2 hours) or 24 hours (plus or minus 2 hours) after the last administration of the study drug at Week 8 or Withdrawal (up to Week 8).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Paroxetine
Number analyzed (Participants) | 18
nanograms per milliliter (ng/mL)
  paroxetine 10 mg, 12 hours, n=4 | 4.4683 (2.16507)
  paroxetine 10 mg, 24 hours, n=3 | 8.9713 (7.81518)
  paroxetine 20 mg, 12 hours, n=1 | 49.5820 (0)
  paroxetine 20 mg, 24 hours, n=3 | 18.2713 (9.78765)
  paroxetine 30 mg, 12 hours, n=2 | 64.4285 (23.34372)
  paroxetine 40 mg, 12 hours, n=3 | 108.9133 (9.01693)
  paroxetine 40 mg, 24 hours, n=2 | 67.9855 (4.08778)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected during the treatment (8 weeks at maximum) and taper phases (3 weeks at maximum). SAEs were also collected during the follow-up phase (2 weeks after the last dose of investigational product).
Arm/Group | Placebo | Paroxetine
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/29
Other Adverse Events (participants affected / at risk) | 9/27 | 9/29
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | Paroxetine (N=29)
Nasopharyngitis (Infections and infestations) | 4 | 6
Influenza (Infections and infestations) | 2 | 1
Suicidal ideation (Psychiatric disorders) | 3 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 1
Headache (Nervous system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.